CLINICAL TRIAL: NCT06418152
Title: Dual-task Augmented Reality Treatment (DART) for Parkinson's Disease and Deep Brain Stimulation
Brief Title: Dual-task Augmented Reality for PD DBS
Acronym: DART for DBS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jay Alberts (Other)
Responsible Party: Sponsor-Investigator, Jay Alberts, Center Director, The Cleveland Clinic
Organization: The Cleveland Clinic (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24-282
Record Dates: First submitted 2024-05-09; First posted 2024-05-17 (Actual); Results first posted 2025-09-30 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Parkinson's Disease; Deep Brain Stimulation
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: 5 to 10 individuals with previously implanted deep brain stimulation and Parkinson's disease
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Interventional Arm (Experimental): Five to ten individuals with PD and DBS will receive the DART intervention. The 16 DART sessions will be delivered over an 8-week period (but not more than 10-weeks). Each DART session will consist of approximately 30-minutes of dual-task activity and will be scheduled over a 1 hour period. A physical therapist or physical therapist assistant will oversee each session. Exercises will be progressed based on results from the DART platform, feedback from the participant, and the clinical expertise of the physical therapist or physical therapist assistant
  Interventions: Behavioral: Multi-modal treatment

INTERVENTIONS:
Behavioral: Multi-modal treatment — Multi-modal treatment was designed to target PD-specific declines in the areas of cognitive function and gait and posture impairments. MMT consists of simultaneously training a motor and cognitive task.

SUMMARY:
The goal of this project is to evaluate the safety and preliminary effectiveness of utilizing a digital therapeutic, Dual-task Augmented Reality Treatment (DART) protocol, for the treatment of postural instability and gait dysfunction (PIGD) in individuals with PD with a previously implanted deep brain stimulator (DBS).

DETAILED DESCRIPTION:
Multi-Modal Training in PD patients: In order to treat dual-task impairment (difficulty performing two tasks at once), multi-modal treatment (MMT) was designed to target PD-specific declines in the areas of cognitive function and gait and posture impairments. Briefly, MMT training consists of simultaneously training a motor and cognitive task. The motor aspect of MMT stresses high velocity, high amplitude training principles while the cognitive aspect stresses commonly impaired cognitive domains in PD such as attention and executive function. An example of an MMT task is marching while spelling words backwards.

Delivery of a Digital Therapeutic via Augmented Reality for the Treatment of PIGD: The MMT intervention is well-suited for integration into an augmented reality (AR) platform as it consists of the patient performing a series of cognitive and motor tasks simultaneously while the patient receives knowledge of performance and results from a therapist. The Microsoft HoloLens is an untethered, AR headset used in applications as broad as teaching anatomy, displaying fine art and gaming. With AR, the user maintains contact with the physical world and the people in it. The HoloLens uses AR technology to place holograms, objects made entirely of projected light, into the user's physical environment; hence creating a first-person mixed reality environment. These holograms can be viewed from different angles and distances, can be two-dimensional or three-dimensional, can appear life-like, can move, be shaped, and change according to interaction with users' or the physical environment in which they are projected, depending on the programming. The MMT was previously developed for the Dual-task Augmented Reality Treatment (DART), which delivers MMT training on a head-mounted AR display. The DART platform was successfully piloted in 50 individuals with PD who did not have DBS (IRB # 20-207). The results of the project indicate that DART is an effective method of training for individuals with PD. The goal is to expand the impact of that project through the investigation of DART in individuals with PD who have previously undergone DBS surgery.

ELIGIBILITY:
Inclusion Criteria:

* Adult with a diagnosis of idiopathic PD
* History of deep brain stimulator placement for treatment of PD
* Ability to ambulate > 10 minutes continuously without an assistive device

Exclusion Criteria:

* Medical diagnosis of dementia or any neurocognitive impairment that compromises the ability to provide informed consent

  ->2 errors on the Short Portable Mental Status Questionnaire
* Musculoskeletal or cardiopulmonary issue that limits one's ability to engage in exercise
* Neurological disease other than Parkinson's disease that impacts motor or cognitive function

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2024-05-21 (Actual); Primary Completion 2025-01-30 (Actual); Study Completion 2025-01-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Cleveland Clinic Foundation, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited beginning May 21, 2024 through December 2024.
Pre-assignment Details: All participants were in the same arm of this pilot study.
Period: Overall Study
Arm/Group | Interventional Arm
Started | 7
Completed | 4
Not Completed | 3
Not completed — Frequent DBS setting changes | 1
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Groups:
- Interventional Arm: Up to five individuals with PD and DBS will receive the DART intervention. The 16 DART sessions will be delivered over an 8-week period (but not more than 10-weeks). Each DART session will consist of approximately 30-minutes of dual-task activity and will be scheduled over a 1 hour period. A physical therapist or physical therapist assistant will oversee each session. Exercises will be progressed based on results from the DART platform, feedback from the participant, and the clinical expertise of the physical therapist or physical therapist assistant
  Multi-modal treatment: Multi-modal treatment was designed to target PD-specific declines in the areas of cognitive function and gait and posture impairments. MMT consists of simultaneously training a motor and cognitive task.
Arm/Group | Interventional Arm
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.5 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 4
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 4
Movement Disorder Society-Unified Parkinson's Disease Rating Scale (Motor Examination) [Mean (Standard Deviation); unit: units on a scale] — Movement Disorder Society Unified Parkinson's Disease Rating Scale Part III: Motor Examination score, measured off medication. Range of scores is 0 to 132, with lower score indicating better motor function.
  units on a scale | 38 (16)

OUTCOME MEASURES:

1. Primary Outcome: Movement Disorder Society Unified Parkinson's Disease Rating Scale Part III: Motor Examination Score
Description: Movement Disorder Society Unified Parkinson's Disease Rating Scale Part III: Motor Examination score, measured off medication. Range of scores is 0 to 132, with lower score indicating better motor function.
  Change in MDS-UPDRS III score from baseline through completion.
Time Frame: Baseline and through study completion, average 8 weeks
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Interventional Arm
Number analyzed (Participants) | 4
Score on a scale | 3.25 (3.27)

2. Secondary Outcome: Two Minute Walk Test
Description: Distance traveled during a 2 minute period under single-and dual-task conditions. Number reported is the change in distance from baseline to end of intervention.
Time Frame: Baseline and through study completion, average 8 weeks
Measure: Mean (Standard Deviation); unit: meters/second
Arm/Group | Interventional Arm
Number analyzed (Participants) | 4
meters/second | 0.06 (0.15)

ADVERSE EVENTS:
Time Frame: Adverse events were collected during active study participation dates. The study intervention from baseline testing to end of testing was an 8-week period, not to exceed 10-weeks. Participants were asked at each session whether any adverse events occurred since the previous session.
Arm/Group | Interventional Arm
All-Cause Mortality (participants affected / at risk) | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 2/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Interventional Arm (N=7)
Non-serious adverse event (Musculoskeletal and connective tissue disorders) | 1 (1) — Back pain, potentially related to study participation
Non-serious adverse event (Injury, poisoning and procedural complications) | 1 (1) — Fall during study intervention.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-11-04): https://cdn.clinicaltrials.gov/large-docs/52/NCT06418152/Prot_SAP_000.pdf